CLINICAL TRIAL: NCT04114136
Title: A Phase II Clinical Trial of Anti-PD-1 mAb Therapy Alone or With Metabolic Modulators to Reverse Tumor Hypoxia and Immune Dysfunction in Solid Tumor Malignancies
Brief Title: Anti-PD-1 mAb Plus Metabolic Modulator in Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dan Zandberg (Other)
Responsible Party: Sponsor-Investigator, Dan Zandberg, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 18-190
Record Dates: First submitted 2019-09-26; First posted 2019-10-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Melanoma; NSCLC; Hepatocellular Carcinoma; Urothelial Cancer; Gastric Adenocarcinoma; HNSCC; Esophageal Adenocarcinoma; Microsatellite Instability-High Solid Malignant Tumor
Keywords: Anti-PD-1 monoclonal antibody (mAb); tumor infiltrating lymphocytes (TIL)
MeSH Terms: conditions — Melanoma; Carcinoma, Hepatocellular; Squamous Cell Carcinoma of Head and Neck; Adenocarcinoma Of Esophagus | interventions — Nivolumab; pembrolizumab; Metformin; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anti-PD-1 mAb (nivolumab or pembrozilumab) plus Metformin (Experimental): nivolumab (480mg IV q 4 weeks) or pembrozilumab (200mg IV q 3 weeks) - dependent upon approved indication. (If both agents are approved for the disease indication, selection is at the discretion of the investigator)
  Metformin - 500 mg by mouth twice daily
  Interventions: Drug: Nivolumab or Pembrolizumab (dependent upon approved indication); Drug: Metformin
- Anti-PD-1 mAb (nivolumab or pembrozilumab) plus Rosiglitazone (Experimental): nivolumab (480mg IV q 4 weeks) or pembrozilumab (200mg IV q 3 weeks) - dependent upon approved indication. (If both agents are approved for the disease indication, selection is at the discretion of the investigator)
  Rosiglitazone - 4 mg by mouth once daily
  Interventions: Drug: Nivolumab or Pembrolizumab (dependent upon approved indication); Drug: Rosiglitazone
- Anti-PD-1 mAb (nivolumab or pembrozilumab) (Active Comparator): nivolumab (480mg IV q 4 weeks) or pembrozilumab (200mg IV q 3 weeks) - dependent upon approved indication. (If both agents are approved for the disease indication, selection is at the discretion of the investigator)
  Interventions: Drug: Nivolumab or Pembrolizumab (dependent upon approved indication)

INTERVENTIONS:
Drug: Nivolumab or Pembrolizumab (dependent upon approved indication) — Anti-PD-1 mAb (monoclonal antibody)
  Other Names: Opdivo (nivolumab) or Keytruda (pembrolizumab)
Drug: Metformin — Acts directly or indirectly on the liver to lower glucose production, and acts on the gut to increase glucose utilisation, increase GLP-1 and alter the microbiome.
  Other Names: Glucophage, Glucophage XR, Fortamet, and Glumetza
  Arms: Anti-PD-1 mAb (nivolumab or pembrozilumab) plus Metformin
Drug: Rosiglitazone — A member of the thiazolidinedione class of antidiabetic agents, improves glycemic control by improving insulin sensitivity. Rosiglitazone is a highly selective and potent agonist for the peroxisome proliferator-activated receptor-gamma (PPARγ).
  Other Names: Avandia
  Arms: Anti-PD-1 mAb (nivolumab or pembrozilumab) plus Rosiglitazone

SUMMARY:
Patients with histologically or cytologically confirmed advanced melanoma, renal cell carcinoma, NSCLC, HCC (Child Pugh Class A only), MSI-High solid tumors, Urothelial Cancer, GE junction/Gastric Adenocarcinoma, or HNSCC for which current standard of care treatment for their stage of disease would be with Pembrolizumab or Nivolumab monotherapy, who meet eligibility criteria will undergo a biopsy (core or excisional/incisional; FNA not adequate) for baseline tissue. Patients will then be randomized to one of 3 arms: Anti-PD-1 mAb plus Metformin 500mg po BID, Anti-PD-1 mAb alone, Anti-PD-1 mAb plus Rosiglitazone 4mg po qdaily. Five weeks (+/- 7 days) after initiation of therapy a patient will undergo a repeat biopsy (core or excisional/incisional; FNA not adequate) for correlative analysis. The patient will then continue on study therapy for up to 2 years, or until progression of disease or unacceptable toxicity, whichever occurs first. RECIST 1.1 with modifications, to allow for continued therapy until progressive disease is confirmed if the patient is clinically stable, will be used in the trial.

DETAILED DESCRIPTION:
The prognosis for patients with metastatic disease remains poor. The use of immunotherapy in the treatment of cancer is based on the premise that tumors evade the endogenous immune response by being recognized as self, and not non-self. The recent success of immune-modulating agents in patients with refractory solid tumors has provided proof-of-concept of the efficacy of immune system activation as a therapeutic modality. Tumors develop immune resistance using different mechanisms; the goal of immunotherapy is to counteract these resistance mechanisms, allowing the endogenous immune system to reject tumors. One of those mechanisms of resistance is tumor hypoxia

This study aims to examine whether Metformin and Rosiglitazone will reduce tumor oxygen consumption, creating a less hypoxic T cell environment, with pharmacologic remodeling of the TME leading to restored anti-tumor T cell effector function and as a result will act synergistically with anti-PD-1 mAb resulting in a higher response rate than with anti-PD-1 mAb alone. The safety and tolerability of if adding metformin or rosiglitazone to anti-PD-1 mAb therapy will assessed.

Eligible patients will undergo pre-treatment biopsy and then will be randomized to one of three arms: 1. Anti-PD-1 mAb + Metformin 500mg PO BID 2. Anti-PD-1 mAb alone or 3. Anti-PD-1 mAb plus Rosiglitazone 4mg po qdaily. Patients will undergo post treatment biopsy after 5 weeks (+/- 7 days) of treatment and then continue treatment for up to 2 years, or until progression of disease or unacceptable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced melanoma, renal cell carcinoma, NSCLC, HCC (Child Pugh Class A only), MSI-High solid tumors, Urothelial Cancer, GE junction/Gastric Adenocarcinoma, or HNSCC for which current standard of care treatment for their stage of disease would be with Pembrolizumab or Nivolumab monotherapy.
2. Accessible tumor for pretreatment (baseline) and post treatment biopsy. Tumor must be accessible for core or surgical biopsy (excisional/incisional), FNA is not adequate
3. Age ≥ 18 years
4. Have at least one measurable area of disease (Target Lesion) based on RECIST 1.1.
5. ECOG performance status 0-2
6. Patients must have normal organ and marrow function as defined below:

   absolute neutrophil count ≥1,500/mcL platelets ≥100,000/mcL total bilirubin ≤ institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN Creatinine clearance ≥40 mL/min/1.73 m2
7. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use one methods of birth control or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Women of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
10. Ability to understand and the willingness to sign a written informed consent document
11. If known to have prior brain metastases, must not have evidence of active (enlarging and/or symptomatic lesions) brain disease on MRI/CT evaluation.
12. A type II DM patient who does not currently require prescription medication for diabetes treatment and has not received metformin, insulin, sulfonylureas or thiazolidinediones within 60 days of the start of study treatment can be enrolled on the study.

Exclusion Criteria:

1. Treatment with prior anti-PD-1 or anti-PD-L1 mAb therapy
2. Patients with type I DM or any patient who has received metformin, insulin, sulfonylureas, or thiazolidinediones within 60 days of start of study treatment for any reason.
3. Pregnancy or breastfeeding. Women of childbearing potential (WOCBP) must practice acceptable methods of birth control to prevent pregnancy. Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study must be informed of the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
4. All WOCBP MUST have a negative pregnancy test within 7 days prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study.
5. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic therapy or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
6. History of uncontrolled cardiac disease (e.g., uncontrolled hypertension, unstable angina, myocardial infarction within prior 6 months)
7. Symptomatic heart failure or New York Heart Association Class III or IV heart failure
8. Psychiatric illness or other social issues limiting compliance
9. Has a history of non-infectious pneumonitis that required steroids, evidence of interstitial lung disease, or currently active non-infectious pneumonitis.
10. Treatment with a non-approved or investigational drug within 14 days prior to Day 1 of study treatment.
11. Prior malignancy within 2 years with the exception of adequately treated basal cell or squamous cell skin cancer, carcinoma of the cervix or prostate cancer.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies). Per Medical History Review
14. Hypersensitivity to metformin, rosiglitazone, pembrolizumab or nivolumab
15. Unable to take in pills either orally or via feeding tube
16. History of acidosis of any type or habitual intake of 5 or more alcoholic beverages a day.
17. Patients that require active treatment with Rifampin or Gemfibrozil for other medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2032-04-30 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Best overall response | From start of the treatment until disease progression/recurrence up to 48 months
  Best overall response per Response Evaluation Criteria in Solid Tumors (RECIST v1.1), by tumor type, recorded from the start of the treatment until disease progression/recurrence. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or non-target) with reduction in short axis to <10 mm. Partial Response (PR): ≥ 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Incomplete Response/Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, (reference smallest sum diameters). Progressive Disease (PD): ≥ 20% increase in the sum of diameters of target lesions (reference smallest sum diameters); the sum must also demonstrate an absolute increase of at least 5 mm; (appearance ≥ 1 new lesions is considered progression).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 48 months
  The length of time after study enrollment that patients lives without experiencing disease progression per RECIST v1.1. Progressive Disease (PD): ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Overall Survival (OS) | Up to 48 months
  The length of time after study enrollment that patients remain alive.
Number of Participants Experiencing Adverse Events Attributed to Treatment | Up to 48 months
  Participants experiencing adverse events (per CTCAE v5.0) that are possibly, probably or definitely related to study treatment, will be tabulated by category, grade and relatedness.

OTHER OUTCOMES:
Change in Lymphocyte Cell Status | Up to 48 months
  Percent of T cell proliferation (increase in number of cells) in peripheral blood prior to treatment compared to post treatment. T cell proliferation is associated with anti-tumor response.
Restoration (change) of Mitochondrial Function in Nodal Infiltrating Lymphocytes | Up to 48 months
  Percent of mitochondrial restoration in nodal infiltrating lymphocytes (located within tumor) prior to treatment compared to post treatment. Functional mitochondria might ultimately lead to the restoration of apoptosis in cancer cells that are refractory to current anticancer agents.
Restoration (change) of Mitochondrial Function in Peripheral Blood Lymphocytes | Up to 48 months
  Percent of mitochondria restoration in peripheral blood lymphocytes prior to treatment compared to after treatment. Functional mitochondria might ultimately lead to the restoration of apoptosis in cancer cells that are refractory to current anticancer agents.

CONTACTS AND LOCATIONS:
Overall Officials: Dan P Zandberg, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zandberg DP, Menk AV, Velez M, Normolle D, DePeaux K, Liu A, Ferris RL, Delgoffe GM. Tumor hypoxia is associated with resistance to PD-1 blockade in squamous cell carcinoma of the head and neck. J Immunother Cancer. 2021 May;9(5):e002088. doi: 10.1136/jitc-2020-002088. PMID 33986123